CLINICAL TRIAL: NCT00734864
Title: Phase I Study of Dasatinib Plus Protracted Temozolomide in Recurrent Malignant Glioma
Brief Title: Ph. I Dasatinib/Protracted Temozolomide in Recurrent Malignant Glioma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug supplier withdrew support for the study. Study was withdrawn from the Duke IRB.
Sponsor: Annick Desjardins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assist Professor of Medicine-Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007909; BMS Protocol #CA180-108
Record Dates: First submitted 2008-05-04; First posted 2008-08-14 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Glioma
Keywords: Dasatinib; Sprycel; Temozolomide; Temodar; Recurrent Malignant Glioma; Malignant Glioma; glioblastoma multiforme; gliosarcoma; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic mixed glioma; glioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Subjects taking EIAEDs (CYP3A enzyme-inducing anti-epileptic drugs).
  Interventions: Drug: enzyme-inducing anti-epileptic drugs
- 2 (Other): Subjects NOT taking EIAEDs (CYP3A enzyme-inducing anti-epileptic drugs).
  Interventions: Drug: enzyme-inducing anti-epileptic drugs

INTERVENTIONS:
Drug: enzyme-inducing anti-epileptic drugs — Subjects taking EIAEDs (CYP3A enzyme-inducing anti-epileptic drugs Phenytoin/Dilantin, Fosphenytoin/Cerebyx, Phenobarbital, Primidone/Mysoline, Oxcarbazepine/Trileptal, Carbamazepine/Tegretol).
  Arms: 1
Drug: enzyme-inducing anti-epileptic drugs — Subjects NOT taking EIAEDs (CYP-3A enzyme-inducing anti-epileptic drugs Phenytoin/Dilantin, Fosphenytoin/Cerebyx, Phenobarbital, Primidone/Mysoline, Oxcarbazepine/Trileptal, Carbamazepine/Tegretol).
  Arms: 2

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of dasatinib when combined with protracted, daily temozolomide (TMZ). Secondary objectives are: To further evaluate the safety and tolerability of dasatinib plus protracted, daily TMZ; 2. To evaluate the pharmacokinetics of dasatinib when administered with protracted, daily TMZ among recurrent malignant glioma patients who are on and not on CYP-3A enzyme inducing anti-epileptic drugs (EIAEDs); 3. To evaluate for anti-tumor activity with this regimen in this patient population.

DETAILED DESCRIPTION:
This is an open-label, single center, one-arm phase I dose-escalation study of dasatinib plus protracted , daily TMZ administered orally on a continuous daily dosing schedule among adult patients with recurrent or relapsing malignant glioma. The study format includes a classical "3+3" dose escalation design to determine the MTD and DLT of dasatinib plus protracted, daily TMZ among recurrent malignant glioma patients. Patients will be stratified based on whether they are receiving EIAED and each stratum will independently dose escalate. Additionally, the study will characterize the safety, tolerability, biologic activity, and pharmacokinetic profile of dasatinib when used in combination with protracted, daily TMZ.

Patients will start treatment on day 1 of cycle 1 with dasatinib. For patients undergoing dasatinib pharmacokinetic (PK) analysis, dasatinib will be administered alone until initial PK assessments are collected. Protracted TMZ will be initiated after initial dasatinib PK assessments are collected and will continue to be administered with dasatinib on a continuous daily dosing schedule. The initial dasatinib PK assessments will be collected over 24 hours between days 3-7 of cycle 1. Patients not undergoing dasatinib PK collections will begin both dasatinib and protracted, daily TMZ together on day 1, cycle 1.

The protracted, daily TMZ dose will be 50 mg/m² daily for all patients. The dose level of dasatinib will be increased in successive cohorts. Cohorts of 3-6 patients will accrue at each dose level until MTD is defined. Each cohort will consist of a minimum of 3 newly enrolled patients. Intra-patient dose escalation is not permitted. It is estimated that this study will enroll a minimum of 30 patients (up to 4 dose levels/stratum; 3 patients/dose level for levels 1-3 and 6 patients at level 4) and a maximum of 48 patients (6 patients/dose level; 4 dose levels/stratum). Cohorts may be expanded at any dose level for further elaboration of safety and pharmacokinetic parameters as required.

The primary safety and efficacy analysis will be conducted on all patient data at the time all patients who are still receiving study drug will have completed at least 4 cycles of treatment. The additional data for any patients continuing to receive study drug past this time, as allowed by the protocol, will be further summarized in a report once these patients either completed or discontinued the study. Prior to the primary analysis, an additional safety report may be prepared.

The most common side effects include vomiting, diarrhea, anorexia (loss of appetite), fluid retention, fatigue, headache, rash, hypocalcemia (low calcium level), and decreases in blood counts. Other possible side effects may include nausea, joint pain, muscle aches, generalized pain, abdominal pain, and fever. Rare side effects may include QTc prolongation (heart beat changes), pulmonary edema (fluid around the lungs), difficulty breathing, cough, hemorrhage, gastrointestinal bleeding, pneumonia, cardiac effusion (fluid in the sac surrounding the heart), and cardiac failure. Temodar has been well tolerated by both adults and children with the most common toxicity being mild myelosuppression. Other, less likely, potential toxicities include nausea and vomiting, constipation, headache, alopecia, rash, burning sensation of skin, esophagitis, pain, diarrhea, lethargy, hepatotoxicity, anorexia, fatigue and hyperglycemia. As in the case with many anti-cancer drugs, Temodar may be carcinogenic. Rats given Temodar have developed breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed diagnosis of a recurrent/progressive WHO Gr.4 malignant glioma (glioblastoma multiforme or gliosarcoma) or WHO Gr.3 malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or anaplastic mixed glioma). Recurrence will be defined based on the modified MacDonald criteria or based on histopathologic confirmation of tissue obtained via surgical intervention. Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO Gr.III or IV malignant glioma;
2. > or = to 18 y/o;
3. KPS . or = to 60%;
4. Patients must be presenting in 1st, 2nd or 3rd relapse. Relapse is defined as progression following anti-cancer therapy other than surgery, including non-surgical therapies that are considered standard treatment for high-grade glioma if administered to patients with prior low-grade glioma. Prior therapy must have included external beam radiotherapy;
5. Adequate bone marrow, liver and renal function as assessed by the following: Hematocrit > or = to 29%, ANC > or = to 1,500/mm3, Platelet count > or = to 125,000/mm3, Total bilirubin < or = to 1.5 x ULN, ALT and AST < or = to 2.5 x the ULN ( < or = to 5 x ULN for patients with liver involvement), INR < 1.5 or a PT/PTT within normal limits (unless on therapeutic anti-coagulation). Patients receiving anti-coagulation treatment with a low-molecular weight heparin will be allowed to participate, however oral warfarin is not permitted except for low-dose warfarin (1mg po DAILY), Creatinine < 1.5 x ULN, Serum Na, K+, Mg2+, Phosphate and Ca2+ > or = to Lower Limit of Normal (LLN);
6. An interval of at least 2 weeks between prior surgical resection (1 week for biopsy) and initiation of study regimen;
7. An interval of at least 12 weeks from completion of standard, daily XRT, unless one of the following occurs: a) new area of enhancement on MRI imaging that is outside the XRT field; b) biopsy proven recurrent tumor; c) radiographic evidence of progressive tumor on 2 consecutive scans at least 4 weeks apart;
8. An interval of at least 4 weeks from prior chemotherapy (except nitrosoureas which require 6 weeks) unless there is unequivocal evidence of tumor progression and the patient has recovered from all anticipated toxicities from prior therapy;
9. An interval of a least 14 days from exposure to investigational agents, unless there is unequivocal evidence of tumor progression and the patients has recovered from all anticipated toxicities from prior therapy;
10. Signed written informed consent including HIPAA according to institutional guidelines. A signed informed consent must be obtained prior to any study specific procedures;
11. If sexually active, patients will take contraceptive measures for the duration of the treatments and for 3 months following discontinuation of dasatinib and TMZ;
12. Women of childbearing potential must have a negative serum or urine pregnancy test (sensitivity < or = to 25IU HCG/L) within 72 hours prior to the start of study drug administration.

Exclusion Criteria:

1. Prior dasatinib. Imatinib mesylate in the prior three months;
2. Grade 3 or greater toxicity related to prior TMZ therapy;
3. Prior progression on protracted daily TMZ;
4. Pregnancy or breast feeding;
5. History of significant concurrent illness;
6. More than 3 prior episodes of progressive disease;
7. Significant cardiac disease including any of the following:

   1. congestive heart failure > class II NYHA;
   2. unstable angina (anginal symptoms at rest);
   3. new onset angina (began within the last 3 months);
   4. myocardial infarction within the past 6 months;
   5. any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
   6. uncontrolled congestive heart failure; diagnosed congenital long QT syndrome; prolonged QTc interval on pre-entry electrocardiogram (> 450 msec);
8. Excessive risk of bleeding as defined by stroke within the prior 6 months, history of CNS or intraocular bleed, or septic endocarditis;
9. Female patients who are pregnant or breastfeeding, or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to administration of study regimen). Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy;
10. Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study such as pleural or pericardial effusion of any grade, uncontrolled diabetes, uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management), active clinically serious infection > CTCAE Gr.2, history of clinically significant bleeding diathesis or coagulopathy including platelet function disorder (e.g. known von Willebrand's disease) or acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies), impairment of GI function or GI disease that may significantly alter the absorption of the study regimen (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets), ongoing or recent (< or = to 3 months) significant gastrointestinal bleeding;
11. Thrombolic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months;
12. Any hemorrhage/bleeding event > CTCAE Gr.3 within 4 weeks of 1st dose of study drug;
13. Serious non-healing wound, ulcer, or bone fracture;
14. Major surgery, open biopsy or significant traumatic injury within 4 weeks of 1st study drug;
15. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C;
16. Patient is < 3 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed;
17. Patient unwilling to or unable to comply with the protocol including ability to swallow whole pills or presence of any malabsorption syndrome;
18. Concurrent administration of warfarin, rifampin or St. John's Wort, except for low-dose warfarin (1mg po DAILY);
19. Clinically serious infection requiring active intervention (CTCAE Gr.2 or greater);
20. Hypokalemia or hypomagnesemia if it cannot be corrected;
21. Concomitant Medications, consider the following prohibitions:

    1. Drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)

       1. quinidine, procainamide, disopyramide
       2. amiodarone, sotalol, ibutilide, dofetilide
       3. erythromycin, clarithromycin
       4. chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
       5. cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
    2. Drugs that reduce dasatinib exposure such as H2 blockers or proton-pump inhibitors (eg famotidine and omeprazole), which can cause long-term suppression of gastric acid secretion. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is in general not recommended and antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy. However, given that nearly all recurrent malignant brain tumor patients are on dexamethasone for increased intracranial pressure, such patients must also receive effective medical therapy to prevent complications related to increased gastric acid secretion due to chronic dexamethasone therapy. Therefore all patients enrolled on the current protocol will receive standard H2 blocker (preferred) or proton pump inhibitor (PPI) therapy to be administered on a daily basis each evening. Dasatinib will be administered each morning in order to maximize the time interval from administered H2 blocker (preferred) or proton pump inhibitor (PPI).
    3. Drugs that cause hypocalcemia (i.e. IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia).
    4. Any prohibited CYP3A4 inhibitors; 22. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Toxicity assessed using CTCAE v.3.0 | weekly

SECONDARY OUTCOMES:
Progression free and overall survival | continuous
Radiographic response (modified MacDonald Criteria) | every 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: Duke University Medical Center Clinical Trials — http://www.dukehealth.org/clinicaltrials
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/